CLINICAL TRIAL: NCT06963632
Title: A Real-world Study on Golidocitinib-based Therapeutic Regimens for the Treatment of Patients With Peripheral T-cell Lymphoma
Acronym: JOYCE
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, M.D. and Ph.D, Ruijin Hospital
Other Study IDs: golidocitinib-based treatment
Record Dates: First submitted 2025-04-23; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Peripheral T-cell Lymphoma (PTCL)
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First line treatment cohort
- Maintenance treatment cohort
- Salvage treatment cohort

SUMMARY:
This real-world study aims to evaluate the safety and efficacy of golidocitinib-based treatment regimens in patients with peripheral T-cell lymphoma (PTCL), without intervention in the selection of therapeutic strategies. A total of 1,000 PTCL patients are planned to be enrolled. After screening, eligible participants meeting the inclusion and exclusion criteria will be assigned to one of three predefined cohorts:

Cohort 1: Treatment-naïve patients with PTCL or NK/T-cell lymphoma.

Cohort 2: Patients receiving maintenance therapy following remission after first-line induction treatment for PTCL.

Cohort 3: Patients with relapsed or refractory PTCL or relapsed/refractory NK/T-cell lymphoma.

There is no cap on the number of participants in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign and acknowledge understanding of the Informed Consent Form
2. Clinically confirmed diagnosis of peripheral T-cell lymphoma
3. Inclusion of PTCL patients who initiated a Golidocitinib-based treatment regimen within the past 3 months
4. Compliance with clinical management and provision of disease-related historical medical information required for the study, including but not limited to medical records, treatment history, and prior/prescribed therapeutic regimens

Exclusion Criteria:

1. Poor patient adherence
2. Investigator-deemed ineligibility for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral T-cell lymphoma who would benefit from golicitinib
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 24 weeks after enrollment
  Percentage of participants with complete or partial response was determined on the basis of investigator assessments according to 2014 Lugano criteria during the treatment
Safety such as adverse events | up to 4 weeks after the last dose
  Rate of adverse events (AEs)/ serious adverse events (SAEs) in patients with lymphoma receiving Golidocitinib therapy

SECONDARY OUTCOMES:
Duration of Response | Baseline up to data cut-off(up to approximately 3 years)
  Applicable to complete or partial response participants. DoR was defined as the time from the first documented date of complete or partial response until the date of the disease progression or death from any causes.
Progression-free survival | Baseline up to data cut-off(up to approximately 3 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off(up to approximately 3 years)
  Percentage of participants with complete or partial response was determined on the basis of investigator assessments according to 2014 Lugano criteria.

IPD SHARING:
Plan to Share IPD: No